CLINICAL TRIAL: NCT00729482
Title: A Phase II Study of RAD001 (Everolimus) in Patients With Fluoropyrimidine and Platinum-refractory Advanced Gastric Cancer
Brief Title: RAD001 (Everolimus) Salvage Monotherapy in Advanced Gastric Cancer (AGC) Who Failed Standard First-line Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC0801
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Results first posted 2014-02-13 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Stomach Neoplasm
Keywords: RAD001 (everolimus); second-line treatment; advanced gastric cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Treatment Arm (RAD001)
  Interventions: Drug: RAD001

INTERVENTIONS:
Drug: RAD001 — RAD001 (everolimus) 10mg daily administration orally until disease progression and/or intolerability
  Other Names: everolimus

SUMMARY:
This is a phase II study to evaluate RAD001 (Everolimus) in terms of 4-month progression-free survival rate (primary end-point) and response rate, toxicity, and overall survival (secondary end-points) in patients with metastatic and/or advanced inoperable gastric cancer.

Eligibility criteria include histologically proven gastric/gastroesophageal junction cancer who failed previous first-line standard treatment with fluoropyrimidine and platinum-based chemotherapy.

Oral RAD001 (everolimus) 10mg daily will be administered and the dose will be adjusted according to the observed clinical toxicities. Treatment will be continued until disease progression or patient's intolerability to the study drug.

Total of 54 patients will be enrolled to decide whether the proportion of patients who are free from progression at 4 months (16 weeks), P, is less that or equal to 0.15 or greater than or equal to 0.30 to assess the treatment outcome in 48 patients assuming drop-out rate, 10%.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented stomach adenocarcinoma including adenocarcinoma of the esophagogastric junction
* Patients must have non-resectable disease by metastasis or recurrent disease after curative surgical resection with uni-dimensionally measurable disease (at least longest diameter 1 cm on computed tomography scan, or at least 2 cm on chest x-ray or physical examination)
* Patients tumor should have failure of 1st line chemotherapy including fluoropyrimidine (5-FU, capecitabine, doxifluridine, S1, or UFT) and platinum (cisplatin, carboplatin, or oxaliplatin) in palliative setting; progression during or within 6 months after chemotherapy
* Age 18 to 75 years old
* Estimated life expectancy of more than 3 months
* ECOG performance status of 2 or lower
* Adequate bone marrow function
* Adequate kidney function
* Adequate liver function
* No prior radiation therapy to more than 25 percent of BM
* Patients must not have psychological, familial, sociological or geographical conditions which do not permit medical follow-up and compliance with this study
* Women of childbearing potential must have a negative pregnancy test on admission
* The patient must be able to understand the study and has given written informed consent to participate in the study

Exclusion Criteria:

* Other tumor types than adenocarcinoma
* Central nervous system metastases or prior radiation for CNS metastasis
* Gastric outlet obstruction or intestinal obstruction
* Evidence of active gastrointestinal bleeding
* Bony metastasis as the sole evaluable disease
* Past or concurrent history of neoplasm other than stomach cancer
* Pregnant or lactating women, women of childbearing potential not employing adequate contraception
* Thyroid disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-07; Primary Completion 2011-09 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa, South Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- RAD001: Treatment Arm (RAD001) take RAD001 10mg/day dose (two 5mg tablets) orally evert day with a glass of water at the same time each day in a fasting state or with a light fat-free meal.
Period: Overall Study
Arm/Group | RAD001
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis was based on all enrolled patients.
Groups:
- RAD001: Treatment Arm (RAD001)
Arm/Group | RAD001
Number analyzed (Participants) | 54
Age, Customized [Median (Full Range); unit: years] | 57.5 [27 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 45
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 54

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Rate at 4-month (16 Weeks)
Description: progression is definced as a more than 20% increase in one or more lesions or the appearance of any new lesion
Time Frame: 4 months (16 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | RAD001
Number analyzed (Participants) | 54
percentage of participants | 18.4

2. Secondary Outcome: Response Rate
Description: Tumor response is evaluated according to the new guidelines by RECIST criteria (See Appendix D). A complete response (CR) is defined as the disappearance of all evidence of cancer for 4 weeks or longer. A partial response (PR) is defined as a 30% or more reduction in the sum of the longest diameters of target lesions for 4 weeks or longer without any evidence of new lesions or progression of any lesions. Stable disease is defined as less than a 30% reduction or less than a 20% increase in the longest diameters of target lesions without any evidence of new lesions. Progressive disease is defined as a more than 20% increase in one or more lesions or the appearance of any new lesion.
Time Frame: 2years
Population: 51 patients were available for response assessments.
Measure: Number; unit: percentage of participants
Arm/Group | RAD001
Number analyzed (Participants) | 51
percentage of participants | 3.7

3. Secondary Outcome: Overall Survival
Time Frame: 1 year
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | RAD001
Number analyzed (Participants) | 54
Months | 8.3 [4.5 to 12.1]

4. Secondary Outcome: Number of Participants With Adverse Events
Description: (according to National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0)
Time Frame: up to 24 weeks
Measure: Number; unit: participants
Arm/Group | RAD001
Number analyzed (Participants) | 54
participants | 54

ADVERSE EVENTS:
Time Frame: At least 6 months after last dose of chemotherapy.
Arm/Group | RAD001
Serious Adverse Events (participants affected / at risk) | 5/54
Other Adverse Events (participants affected / at risk) | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=54)
Ileus (Gastrointestinal disorders) | 1 — Grade 2 paralytic intestinal obstruction
Pneumonia (Infections and infestations) | 3
Sudden death (Cardiac disorders) | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAD001 (N=54)
Neutropenia (Blood and lymphatic system disorders) | 23
Anemia (Blood and lymphatic system disorders) | 51
Thrombocytopenia (Blood and lymphatic system disorders) | 47
Hypercholesterolemia (Metabolism and nutrition disorders) | 24
Triacylglyceridemia (Metabolism and nutrition disorders) | 13
Hyperglycemia (Metabolism and nutrition disorders) | 47
Hyperbilirubinemia (Hepatobiliary disorders) | 14
Elevated alkaline phosphatase (Hepatobiliary disorders) | 18
Elevated aspartate aminotransferase (Hepatobiliary disorders) | 32
Elevated alanine aminotransferase (Hepatobiliary disorders) | 20
Elevated gamma glutamyl transpeptidase (Hepatobiliary disorders) | 17
Hypophosphatemia (Metabolism and nutrition disorders) | 14
Hyponatremia (Renal and urinary disorders) | 24
Asthenia (General disorders) | 52
Myalgia (Musculoskeletal and connective tissue disorders) | 20
Diarrhea (Gastrointestinal disorders) | 19
Constipation (Gastrointestinal disorders) | 15
Anorexia (Gastrointestinal disorders) | 43
Nausea (Gastrointestinal disorders) | 21
Stomatitis (Gastrointestinal disorders) | 41
Skin rash (Skin and subcutaneous tissue disorders) | 35
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 13
Hemorrhage (Blood and lymphatic system disorders) | 18
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No